CLINICAL TRIAL: NCT06059820
Title: Prospective Cohort Study of the Effectiveness of Conservative Treatment in Patients With AOSpine Type A2 and A3 Fractures of the Thoracic and Lumbar Spine Without Neurological Deficit
Brief Title: Effectiveness of Conservative Treatment in Patients With Thoracic and Lumbar Fractures Without Neurological Deficit
Status: Completed | Type: Observational
Sponsor: Sklifosovsky Institute of Emergency Care (Other Government)
Responsible Party: Principal Investigator, Ivan Lvov, MD, PhD, neurosurgeon, Sklifosovsky Institute of Emergency Care
Other Study IDs: 1-28-08/2023
Record Dates: First submitted 2023-09-22; First posted 2023-09-29 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Thoracic Spine Fracture; Lumbar; Spine, Fracture; Thoracolumbar Burst Fracture; Fracture of Spine, Level Unspecified; Spine Fusion; Spine Fracture
Keywords: Thoracic Spine Fracture; Lumbar Spine Fracture; thoracolumbar burst; Spine fusion; conservative treatment for spine fracture
MeSH Terms: conditions — Fractures, Bone; Spinal Fractures | interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conservative treatment group: The main group (prospective) will consist of patients who received conservative therapy. The expected number of observations in the main group will be 50 patients.
  Interventions: Other: rehabilitation treatment
- Surgical treatment group: The control group (historical control) will be comprised of 50 patients who underwent surgery previously at the Sklifosovsky Research Institute for Emergency Medicine.
  Interventions: Procedure: Spine fusion

INTERVENTIONS:
Other: rehabilitation treatment — 3-month immobilization period, hyperextension braces for specific fractures, therapeutic exercises, and gradual activity restoration.
  Groups: Conservative treatment group
Procedure: Spine fusion — Pedicle screw fixation or fusion; anterior plate fusion
  Groups: Surgical treatment group

SUMMARY:
The goal of this observational study is to compare the long-term clinical outcomes of two treatment methods (conservative therapy and surgical treatment) in patients with fractures of the thoracic and lumbar spine without neurological deficit

DETAILED DESCRIPTION:
The main objectives of the upcoming study include:

* to conduct a retrospective analysis of the surgical treatment outcomes in patients with thoracic or lumbar vertebral fractures;
* to assess the immediate and long-term outcomes of conservative therapy in patients with thoracic or lumbar vertebral injuries;
* to evaluate the overall cost of surgical and conservative treatment one year post-discharge, as well as the duration of disability in patients with thoracic or lumbar vertebral fractures;
* to compare the results of surgical and conservative treatment methods in patients with thoracic or lumbar vertebral fractures.

The research focus will be on patients diagnosed with uncomplicated fractures of the thoracic and lumbar spine, classified as type A2 and A3 according to the AOSpine classification.

Two patient groups will be formed:

The main group (prospective) will consist of patients who underwent conservative therapy. The expected number of observations in the main group will be 40 patients.

The control group (historical control) will be comprised of 40 patients who underwent surgery previously at the Sklifosovsky Research Institute for Emergency Medicine.

The first stage of conservative therapy will be administered within 7 days at the departments of the Sklifosovsky Research Institute for Emergency Medicine. Subsequently, the patient will be transferred to a rehabilitation center for the second stage of conservative treatment at Branch No. 3 of the State Autonomous Healthcare Institution "Moscow Scientific and Practical Center for Medical Rehabilitation, Restorative and Sports Medicine". The third stage of medical rehabilitation will be carried out at outpatient healthcare facilities based on the patient's place of residence.

The study will be considered complete when the data from the final examination of at least 50 patients in each group have been analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 65 years.
* Isolated fracture of a single thoracic or lumbar vertebra, classified as type A2 or A3 according to the AOSpine classification.
* Absence of clinical evidence of nerve root or spinal cord compression at the injury level.
* Degree of spinal canal space narrowing less than 50% based on CT scans.
* Informed consent to participate in the study.

Exclusion Criteria:

* Sagittal imbalance (Type 4 by C. Barrey).
* Vertebral bone density at the injury level less than 100 HU or osteoporosis exceeding grade 3 in vertebral bodies, pelvic bones, and limbs.
* Previous spinal surgeries.
* Anesthesia risk of 4 or 5 according to ASA.
* Acute exacerbation and decompensation of somatic diseases.
* Malignant tumors at any site.
* Systemic connective tissue disorders.
* Cognitive impairments hindering patient communication.
* Floating and mural thrombosis, regardless of location.
* Newly identified and uncorrectable cardiac rhythm disorders.
* Dizziness.
* Consequences of a previous acute cerebrovascular event.
* Pregnancy at any stage.
* Acute infectious diseases.
* History of fractures of the pelvis, lower limbs, or vertebral bodies.
* Congenital spinal and limb disorders.
* Any conditions contraindicating physiotherapeutic procedures.
* Patient refusal to participate in the study.
* Inability to participate in follow-up examinations for one year after the injury.
* Participation in other clinical trials.
* Absence of a signed informed voluntary consent for medical interventions and processing of personal data or personal data processing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants in the study are patients with spinal fractures who arrived through the emergency medical services and were urgently admitted to the hospital.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-09-29 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index | admission, 3, 6 and 12 months
  This questionnaire allows for a precise numeric assessment of the extent to which an individual's daily functioning is affected by back pain and objectively demonstrates the clinical outcome of the provided treatment. The scale will be applied at all stages of the study, starting from the initial examination and concluding with the follow-up examination one year after intervention. The questionnaire consists of 10 sections, each containing 6 statements. Depending on the response, a score from 0 to 5 is assigned. The maximum total score is 50. Subsequently, the scores are converted into percentages, ranging from 0 to 100%. If one of the sections is not applicable or omitted for ethical reasons, the sum of scores from the remaining 9 sections is divided by 45 to calculate the percentage.

SECONDARY OUTCOMES:
The SF-36 v.1 (Standard Form) | admission, 3, 6 and 12 months
  This questionnaire allows for a comprehensive assessment of the quality of life. The questionnaire consists of 36 questions grouped into 8 scales, evaluating physical functioning, role limitations, bodily pain, general health, vitality, social functioning, emotional well-being, and mental health. Each scale has a maximum score of 100 points.
EQ-5D-5L | admission, 3, 6 and 12 months
  This scale is similar to the SF-36 but provides a less detailed assessment of the social adaptation of patients and their emotional well-being. Nevertheless, this questionnaire is frequently used in prospective international research studies. Therefore, we consider it practical to use it to preserve the option for comparative analysis of our results with literature data. The questionnaire consists of 5 sections (mobility, self-care, usual activities, pain, anxiety), each with three statements, and a visual analogue scale EQ-VAS. The results can be converted into a single numerical value (index) adjusted for the patient's region of residence. Currently, there is no complete set of values to calculate this index for the Russian Federation, so in the initial stages, simple comparison of specific numerical values for each parameter will be used. When the technical capability becomes available, the index will be calculated at the end of the study.
ASA | admission
  This classification categorizes patients into 5 classes based on the presence of comorbid conditions (Class I - healthy patient, Class V - moribund patient).
Rivermead Mobility Index | 1, 3, 6 and 12 months
  The Rivermead Mobility Index (RMI) is a tool used to assess the mobility of patients, particularly after injuries or conditions such as stroke. This index is designed to measure a patient's ability to perform various motor tasks and includes an evaluation of aspects such as getting out of bed, moving around a room, descending stairs, and other mobility skills.
  The Rivermead Mobility Index consists of several questions and items, each of which is assigned a specific score. All scores are then summed to determine the overall mobility index. This tool can be used for both medical and research purposes to assess patients' physical function and mobility.
Lovett's muscle testing | 1, 3, 6 and 12 months
  Lovett's method is a clinical technique to assess erector spinae muscle strength. It involves having the patient perform specific movements or resist against applied force. This evaluates muscle strength and functional status. It's used in medical and physical therapy assessments for the lower back.

CONTACTS AND LOCATIONS:
Overall Officials: Andrey Grin, MD, PhD, Study Chair — Sklifosovsky Research Institute for Emergency Medicine; Aleksandr Talypov, MD, PhD, Study Director — Sklifosovsky Research Institute for Emergency Medicine; Vasiliy Karanadze, MD, PhD, Principal Investigator — Sklifosovsky Research Institute for Emergency Medicine; Ivan Lvov, MD, PhD, Principal Investigator — Sklifosovsky Research Institute for Emergency Medicine; Anton Kordonskiy, MD, PhD, Principal Investigator — Sklifosovsky Research Institute for Emergency Medicine; Iren Pogonchenkova, MD, PhD, Study Chair — Moscow Scientific and Practical Center for Medical Rehabilitation, Restorative and Sports Medicine
Locations (2):
- Russia (2):
  - Sklifosovsky Research Institute for Emergency Medicine, Moscow
  - Moscow Scientific and Practical Center for Medical Rehabilitation, Restorative and Sports Medicine, Moscow

IPD SHARING:
Plan to Share IPD: Yes
All the obtained data will be stored in the data centre of the Sklifosovsky Research Institute for Emergency Medicine. These data will be unavailable to all parties until the final analysis.
Supporting Information: Study Protocol, SAP, ICF, CSR